CLINICAL TRIAL: NCT04879511
Title: Effect of Metformin on Circulating Neuregulin-4 in Children With Type 1 Diabetes
Brief Title: Effect of Metformin in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nancy Samir Elbarbary, Prof.of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ain shams Pediatrics 2102018
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Effect of Change in T1DM Glycemic Control
Keywords: Neuregulin-4; metformin; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Receiving metformin (Active Comparator): Active group receiving metformin with basal /bolus insulin
  Interventions: Drug: metformin; Drug: Basal/bolus insulin
- Placebo (Placebo Comparator): Control group receiving Placebo with basal/bolus insulin
  Interventions: Drug: Basal/bolus insulin

INTERVENTIONS:
Drug: metformin — Oral hypoglycemic drug metformin
  Other Names: Glucophage
  Arms: Receiving metformin
Drug: Basal/bolus insulin — Basal/bolus insulin

SUMMARY:
Cardiovascular disease is the leading cause of mortality in type 1 diabetes mellitus (T1DM). Vascular dysfunction is an early and critical event in the development of cardiovascular disease. Children with T1DM have vascular dysfunction therefore early interventions to improve vascular health are essential to reduce cardiovascular mortality in T1DM. Metformin is an insulin sensitising agent which is known to improve vascular health outcomes in type 2 diabetes mellitus (T2DM) and other individuals with insulin resistance. It has been used safely in children and adolescents with T2DM for over 10 years. This study aims to assess the effect of metformin on vascular health in children with T1DM.

This is the first study to study effect of metformin on circulating neuregulin-4 levels as a marker for subclinical atherosclerosis.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is an autoimmune disease characterized by T-cell mediated destruction of the pancreatic b-cells, resulting in insulin deficiency and elevated blood glucose levels.

The increasing incidence of type 1 diabetes mellitus in many countries challenges health systems because the disease is presently incurable with no known method of prevention. Around 490,100 children live with the disease worldwide, with incidence estimated to be increasing in children under 15 years by 2.8% per year .This trend is particularly worrying because type 1 diabetes increases mortality and morbidity population-wide.

Vascular co-morbid diseases include retinopathy, which may cause reduced vision and blindness, and nephropathy, which may result in renal failure and require dialysis or kidney transplantation. This is in addition to hypertension, which is linked to peripheral, cardio- and cerebrovascular disease, the end points of which are limb amputations, cardiac failure, stroke and sudden death. As vascular complications curtail both life expectancy and quality of life development at younger ages when people are typically establishing Type 1 diabetes mellitus (T1DM) is an autoimmune disease characterized by T-cell mediated destruction of the pancreatic b-cells, resulting in insulin deficiency and elevated blood glucose levels.

The increasing incidence of type 1 diabetes mellitus in many countries challenges health systems because the disease is presently incurable with no known method of prevention . Around 490,100 children live with the disease worldwide, with incidence estimated to be increasing in children under 15 years by 2.8% per year .This trend is particularly worrying because type 1 diabetes increases mortality and morbidity population-wide.

Vascular co-morbid diseases include retinopathy, which may cause reduced vision and blindness, and nephropathy, which may result in renal failure and require dialysis or kidney transplantation. This is in addition to hypertension, which is linked to peripheral, cardio- and cerebrovascular disease, the end points of which are limb amputations, cardiac failure, stroke and sudden death. As vascular complications curtail both life expectancy and quality of life development at younger ages when people are typically establishing careers and families is particularly detrimental .

Neuregulin 4 (Nrg4), a recently identified adipokine, has been found in multiple organs, in particular brown adipose tissue (BAT), and belongs to the epidermal growth factor (EGF) family of extracellular ligands. Overexpression of Nrg4 can reduce chronic inflammation through inhibiting the gene expression of macrophage marker monocyte chemotactic protein 1 (Mcp1) and enhancing the expression of M2 macrophage marker gene Cd163, demonstrating that Nrg4 may possess anti-inflammatory and anti-atherogenic properties. Lower Nrg4 levels have been reported to be associated with the percentage of body fat mass, liver fat content, obesity, IR, impaired glucose tolerance (IGT), and type 2 diabetes mellitus (T2DM) .

Moreover, serum Nrg4 levels have been reported to be inversely associated with subclinical cardiovascular disease (CVD) in obese adults.

Recent studies reveal that neuregulin.4 may be closely associated with non-alcoholic fatty liver disease (NAFLD) and metabolic syndrome (MetS). Many lines of evidence indicate that inflammation is closely associated with atherosclerosis and plays a crucial role in the development of CVD.

Biguanides sensitize body cells to insulin, which may cause a reduction of atherogenic lipid fractions in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes mellitus (5 years duration at least) and with micro-vascular complications.
* Patients on regular visits to clinic.
* Patients on regular insulin therapy.

Exclusion Criteria:

* Any clinical evidence of infection, hematological diseases, tumors, liver dysfunction, urinary tract disorders, connective tissue disease, or other autoimmune diseases.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Glycemic control(HbA1c%) | up to 24 weeks
  Effect of metformin supplementation on Glycemic control(HbA1c%)

SECONDARY OUTCOMES:
circulating neuregulin-4 level | up to 24 weeks
  Effect of metformin supplementation on level of circulating neuregulin-4

CONTACTS AND LOCATIONS:
Overall Officials: Nancy S Elbarbary, MD.PhD, Principal Investigator — Ain Shams University
Locations (1):
- Nancy Elbarbary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Q, Thompson J, Hu Y, Das A, Lesnefsky EJ. Metformin attenuates ER stress-induced mitochondrial dysfunction. Transl Res. 2017 Dec;190:40-50. doi: 10.1016/j.trsl.2017.09.003. Epub 2017 Sep 28. PMID 29040818
- [Background] Chen LL, Peng MM, Zhang JY, Hu X, Min J, Huang QL, Wan LM. Elevated circulating Neuregulin4 level in patients with diabetes. Diabetes Metab Res Rev. 2017 May;33(4). doi: 10.1002/dmrr.2870. Epub 2016 Dec 27. PMID 27862843
- [Background] Kocak MZ, Aktas G, Erkus E, Yis OM, Duman TT, Atak BM, Savli H. Neuregulin-4 is associated with plasma glucose and increased risk of type 2 diabetes mellitus. Swiss Med Wkly. 2019 Oct 27;149:w20139. doi: 10.4414/smw.2019.20139. eCollection 2019 Oct 21. PMID 31656034